CLINICAL TRIAL: NCT03248479
Title: A Phase 1b Trial of Magrolimab Monotherapy or Magrolimab in Combination With Azacitidine in Patients With Hematological Malignancies
Brief Title: Magrolimab Monotherapy or Magrolimab in Combination With Azacitidine in Participants With Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been discontinued due to futility based on the results of a planned analysis of the ENHANCE trial.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5F9005; 2017-000678-12 (EudraCT Number)
Expanded Access: NCT05627466 (No longer available)
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Hematological Malignancies
Keywords: CD47
MeSH Terms: conditions — Hematologic Neoplasms | interventions — magrolimab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- TN MDS Cohort Higher Risk QW 30 mg/kg (Experimental): Participants who are treatment-naive (TN) with higher risk myelodysplastic syndrome (MDS) will receive 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then weekly (QW) starting Cycle 2 up to end of the study. Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- TN MDS Cohort Higher Risk Q2W 30 mg/kg (Experimental): Participants who are TN with higher risk MDS will receive 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then weekly starting Cycle 2 and given every 2 weeks (Q2W) from Cycle 3 up to end of the study. Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- TN/U AML Cohort: Magrolimab + Azacitidine (Experimental): Participants who are treatment-naive or unfit (TN/U) with acute myeloid leukemia (AML) will receive 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then QW starting Cycle 2 and then given QW and Q2W from Cycle 3 up to end of the study. Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- R/R AML Cohort: Magrolimab + Azacitidine (Experimental): Participants with relapsed/refractory (r/r) AML will receive magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg QW and Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- R/R AML Cohort: Magrolimab (Experimental): Participants with r/r AML will receive magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, Day 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Day 11 and Day 15, 30 mg/kg weekly on Cycle 1 Day 22 through end of Cycle 2, and 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab
- Rollover AML Cohort: Magrolimab (Experimental): Participants may receive the same dose level and schedule (30 mg/kg) (i.e., twice weekly) of magrolimab monotherapy in each cycle (each cycle was of 28 days) as previously received on the Phase 1 AML study (SCI-CD47-002), or may transition to once-weekly dosing in this study at the discretion of the Investigator in each 28-day cycle and with Sponsor approval. Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab
- R/R MDS Cohort: Magrolimab + Azacitidine (Experimental): Participants with r/r MDS will receive magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine (Experimental): Participants with r/r MDS will receive magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Participants will receive azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Participants with r/r MDS who do not have an objective response with magrolimab at the first protocol response assessment can have azacitidine added to magrolimab for subsequent cycles.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- R/R MDS Cohort: Magrolimab (Experimental): Participants with r/r MDS will receive 1 mg/kg magrolimab on Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab
- Low Risk MDS Cohort: Magrolimab + Azacitidine (Experimental): Participants with low risk MDS will receive 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Participants will receive azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg. Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine (Experimental): Participants with low risk MDS will receive 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Participants will receive azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg. Maximum treatment duration was up to 4 years.
  Participants with r/r MDS who do not have an objective response with magrolimab at the first protocol response assessment can have azacitidine added to magrolimab for subsequent cycles.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- Low Risk MDS Cohort: Magrolimab (Experimental): Participants with low risk MDS will receive 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Maximum treatment duration was up to 4 years.
  Interventions: Drug: Magrolimab

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: Hu5F9-G4
Drug: Azacitidine — Administered according to region-specific drug labeling either subcutaneously or intravenously
  Other Names: VIDAZA
  Arms: Low Risk MDS Cohort: Magrolimab + Azacitidine; Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine; R/R AML Cohort: Magrolimab + Azacitidine; R/R MDS Cohort: Magrolimab + Azacitidine; R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine; TN MDS Cohort Higher Risk Q2W 30 mg/kg; TN MDS Cohort Higher Risk QW 30 mg/kg; TN/U AML Cohort: Magrolimab + Azacitidine

SUMMARY:
The primary objectives of this study are:

* To confirm the safety and tolerability of magrolimab monotherapy in a relapsed/refractory (R/R) acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) population, and of magrolimab in combination with azacitidine in previously untreated participants with AML or MDS and participants with R/R AML and MDS
* To evaluate the efficacy of magrolimab monotherapy in R/R AML/MDS, and of magrolimab in combination with azacitidine in previously untreated participants with AML/MDS, or R/R AML/MDS as measured by complete remission (CR) rate for participants with AML and higher-risk MDS, and duration of complete response for participants with AML and higher-risk MDS, and duration of CR for participants with AML and higher-risk MDS
* To evaluate the safety, tolerability, and efficacy of magrolimab monotherapy or combination with azacitidine in low-risk MDS participants as measured by red blood cell (RBC) transfusion independence rate

ELIGIBILITY:
Key Inclusion Criteria:

* Meets the criteria below for the appropriate cohort:

  * Relapsed/Refractory Cohorts: Pathologically confirmed relapsed or refractory (primary refractory and/or relapsed refractory) acute myeloid leukemia (AML) or confirmed intermediate, high, or very high risk myelodysplastic syndromes (MDS) that is relapsed, refractory or intolerant to conventional therapy.
  * Treatment-naive/Unfit Cohorts: Previously untreated individuals with histological confirmation of AML who are ineligible for treatment with a standard cytarabine and anthracycline induction regimen; or previously untreated individuals with intermediate, high, or very high risk MDS. Prior and concurrent therapy with hydroxyurea, oral etoposide, erythroid and/or myeloid growth factors is allowed.
  * Rollover Cohort: Individuals on active magrolimab therapy on the Phase 1 AML (SCI-CD47-002; NCT02678338) trial who are deriving clinical benefit by Investigator assessment.
  * RBC transfusion dependent low risk MDS cohort: Transfusion-dependent MDS individuals who are very low or low risk by Revised International Prognostic Scoring System (IPSS-R) with previous treatment with an erythroid stimulating agent or lenalidomide.
* White blood cell (WBC) count ≤ 20 x 10^3/mcL
* Adequate performance status and hematological, liver, and kidney function.

Key Exclusion Criteria:

* Prior treatment with cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα) targeting agents (with exception of magrolimab for individuals in the Rollover cohort).
* Treatment-naive/Unfit Cohorts Only: Any prior anti-leukemic therapy (excluding hydroxyurea or oral etoposide), prior treatment with hypomethylating agents and/or low dose cytarabine.
* Acute promyelocytic leukemia.
* Known inherited or acquired bleeding disorders.
* Previous allogeneic hematopoietic stem cell transplant within 6 months prior to enrollment, active graft versus host disease (GVHD), or requiring transplant-related immunosuppression.
* Clinical suspicion of active central nervous system (CNS) involvement by leukemia.
* Known active or chronic hepatitis B or C infection or HIV.
* Pregnancy or active breastfeeding.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (27):
- United States (26):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego (UCSD), La Jolla, California
  - UCLA Clinical and Translational Research Center (CTRC), Los Angeles, California
  - Chao Family Comprehensive Cancer Center - UC Irvine Medical Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University Of Miami - Miller School Of Medicine, Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/ Boston Children's Hospital, Boston, Massachusetts
  - Mid America Division, Inc., Kansas City, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Herbert Irving Comprehensive Cancer Center-Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennesssee Oncology - Centennial Clinic Location, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Simmons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of WI Froedtert Hospital, Milwaukee, Wisconsin
- Oxford Centre for Respiratory Medicine Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daver NG, Vyas P, Kambhampati S, Al Malki MM, Larson RA, Asch AS, Mannis G, Chai-Ho W, Tanaka TN, Bradley TJ, Jeyakumar D, Wang ES, Sweet K, Kantarjian HM, Garcia-Manero G, Komrokji R, Xing G, Ramsingh G, Renard C, Zeidner JF, Sallman DA. Tolerability and Efficacy of the Anticluster of Differentiation 47 Antibody Magrolimab Combined With Azacitidine in Patients With Previously Untreated AML: Phase Ib Results. J Clin Oncol. 2023 Nov 1;41(31):4893-4904. doi: 10.1200/JCO.22.02604. Epub 2023 Sep 13. PMID 37703506
- [Background] Sallman DA, Asch AS, Kambhampati S, et al. The first-in-class anti-CD47 antibody magrolimab combined with azacitidine is well tolerated and effective in AML patients: phase 1b results. American Society of Hematology (ASH); 2020 05-08 December. Annual Meeting Virtual.
- [Background] Sallman DA, Asch AS, Al Malki MM, et al. The first-in-class anti-CD47 antibody magrolimab (5F9) in combination with azacitidine is effective in MDS and AML patients: ongoing phase 1b results [Abstract]. American Society of Hematology (ASH); 2019 07-10 December. Orlando, FL.
- [Derived] Sallman DA, Al Malki MM, Asch AS, Wang ES, Jurcic JG, Bradley TJ, Flinn IW, Pollyea DA, Kambhampati S, Tanaka TN, Zeidner JF, Garcia-Manero G, Jeyakumar D, Komrokji R, Lancet J, Kantarjian HM, Gu L, Zhang Y, Tan A, Chao M, O'Hear C, Ramsingh G, Lal I, Vyas P, Daver NG. Magrolimab in Combination With Azacitidine in Patients With Higher-Risk Myelodysplastic Syndromes: Final Results of a Phase Ib Study. J Clin Oncol. 2023 May 20;41(15):2815-2826. doi: 10.1200/JCO.22.01794. Epub 2023 Mar 8. PMID 36888930
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=5F9005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and the United Kingdom. 1 participant with low-risk MDS was accidentally enrolled High-risk MDS group.
Pre-assignment Details: 258 participants were screened.
Groups:
- TN MDS Cohort Higher Risk QW 30 mg/kg: Participants who were treatment-naive (TN) with higher risk myelodysplastic syndrome (MDS) received 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then weekly (QW) starting Cycle 2 up to end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- TN MDS Cohort Higher Risk Q2W 30 mg/kg: Participants who were TN with higher risk MDS received 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then weekly starting Cycle 2 and given every 2 weeks (Q2W) from Cycle 3 up to end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- TN MDS Cohort Low Risk QW 30 mg/kg: Participants who were TN with low risk MDS received 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then QW starting Cycle 2 up to end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- TN/U AML Cohort: Magrolimab + Azacitidine: Participants who were treatment-naive or unfit (TN/U) with acute myeloid leukemia (AML) received 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, and then QW starting Cycle 2 and then given QW and Q2W from Cycle 3 up to end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- R/R AML Cohort: Magrolimab + Azacitidine: Participants with relapsed/refractory (r/r) AML received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/ kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg QW and Q2W starting Cycle 3 and thereafter (each cycle was of 28 days).
  Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- R/R AML Cohort: Magrolimab: Participants with r/r AML received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, Day 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Day 11 and Day 15, 30 mg/kg weekly on Cycle 1 Day 22 through end of Cycle 2, and 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- Rollover AML Cohort: Magrolimab: Participants received the same dose level and schedule (30 mg/kg, twice weekly) of magrolimab monotherapy as previously received on the Phase 1 AML study (SCI-CD47-002), or transitioned to once-weekly dosing in this study at the discretion of the Investigator in each 28-day cycle and with Sponsor approval. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab + Azacitidine: Participants with r/r MDS received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days).
  Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with r/r MDS received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Maximum treatment duration was up to 4 years. Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days).
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles.
- R/R MDS Cohort: Magrolimab: Participants with r/r MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Days 11, 15, 22, through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
- Low Risk MDS Cohort: Magrolimab + Azacitidine: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg. Maximum treatment duration was up to 4 years.
- Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) up to the end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg. Maximum treatment duration was up to 4 years.
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles.
- Low Risk MDS Cohort: Magrolimab: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Maximum treatment duration was up to 4 years.
Period: Overall Study
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN MDS Cohort Low Risk QW 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Started | 32 | 63 | 1 | 87 | 19 | 6 | 1 | 17 | 5 | 10 | 9 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 32 | 63 | 1 | 87 | 19 | 6 | 1 | 17 | 5 | 10 | 9 | 5 | 3
Not completed — Death | 12 | 44 | 1 | 72 | 17 | 6 | 1 | 14 | 3 | 7 | 3 | 1 | 1
Not completed — Study terminated by sponsor | 12 | 15 | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 4 | 0
Not completed — Consent withdrawn | 6 | 3 | 0 | 9 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Not reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received ≥ 1 dose of magrolimab.
Groups:
- R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with r/r MDS received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days).
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles. Maximum treatment duration was up to 4 years.
- Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg.
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles. Maximum treatment duration was up to 4 years.
- Low Risk MDS Cohort: Magrolimab: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day
  1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) up to the end of the study. Maximum treatment duration was up to 4 years.
- Total: Total of all reporting groups
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN MDS Cohort Low Risk QW 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab | Total
Number analyzed (Participants) | 32 | 63 | 1 | 87 | 19 | 6 | 1 | 17 | 5 | 10 | 9 | 5 | 3 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 22 | 0 | 17 | 3 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 58
  >=65 years | 20 | 41 | 1 | 70 | 16 | 6 | 1 | 15 | 5 | 9 | 8 | 5 | 3 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9.1) | 67 (11.6) | 66 (NA) — Standard deviation cannot be calculated for 1 participant. | 71 (10.0) | 73 (7.4) | 77 (6.3) | 79 (NA) — Standard deviation cannot be calculated for 1 participant. | 72 (7.2) | 77 (1.7) | 73 (5.3) | 75 (5.9) | 74 (7.7) | 79 (6.4) | 70 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 1 | 37 | 5 | 3 | 1 | 5 | 4 | 3 | 6 | 1 | 1 | 100
  Male | 23 | 39 | 0 | 50 | 14 | 3 | 0 | 12 | 1 | 7 | 3 | 4 | 2 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 1 | 5 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 17
  Not Hispanic or Latino | 29 | 54 | 0 | 81 | 18 | 6 | 1 | 14 | 5 | 9 | 8 | 5 | 3 | 233
  Unknown or Not Reported | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 11
  White | 31 | 54 | 0 | 75 | 15 | 5 | 1 | 16 | 4 | 10 | 6 | 5 | 3 | 225
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 63 | 1 | 85 | 19 | 6 | 0 | 17 | 5 | 10 | 8 | 5 | 3 | 253
  United Kingdom | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and before the first date of new anti-cancer therapy including stem-cell transplant (SCT) and/or any AEs leading to premature discontinuation of study drug.
Time Frame: Up to 4 years
Population: Safety Analysis Set included all participants who received ≥ 1 dose of magrolimab.
Measure: Number; unit: percentage of participants
Groups:
- Rollover AML Cohort: Magrolimab: Participants received the same dose level and schedule (30 mg/kg, twice weekly) of magrolimab monotherapy as previously received on the Phase 1 AML study (SCI-CD47-002) or transitioned to once-weekly dosing in this study at the discretion of the Investigator in each 28-day cycle and with Sponsor approval. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with r/r MDS received magrolimab 1 mg/kg for Cycle 1 Week 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8, 30 mg/kg on Cycle 1 Days 11, 15 and 22 through end of Cycle 2 and then 30 mg/kg QW in Cycle 2 and then 30 mg/kg Q2W starting Cycle 3 and thereafter (each cycle was of 28 days). Participants received azacitidine 75 mg/m^2 on Days 1 to 7 of each cycle (each cycle was of 28 days). Maximum treatment duration was up to 4 years.
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles.
- Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine: Participants with low risk MDS received 1 mg/kg magrolimab on Cycle 1 Week 1 Day 1; 30 mg/kg on Cycle 1 Days 8, 15 and 22; 60 mg/kg on Day 1 of Cycle 2 and subsequent cycles (each cycle was of 28 days) (each cycle was of 28 days) up to the end of the study. Participants received azacitidine 75 mg/m^2 on Days 1 to 5 of each cycle. For participants who could not tolerate 60 mg/kg dose, the dose of magrolimab was reduced to 45 mg/kg. Maximum treatment duration was up to 4 years.
  Participants with r/r MDS who did not have an objective response with magrolimab at the first protocol response assessment had azacitidine added to magrolimab for subsequent cycles.
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN MDS Cohort Low Risk QW 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 1 | 87 | 19 | 6 | 1 | 17 | 5 | 10 | 9 | 5 | 3
percentage of participants | 100 | 96.8 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Complete Remission (CR) Rate For Participants With AML
Description: The CR rate is the percentage of participants who achieved CR without minimal residual disease (CRMRD-), and CR as per European Leukemia Net (ELN) AML recommendations. CRMRD- per ELN was defined as neutrophils ≥1.0 × 10^9/L; platelets ≥100 × 10^9/L and <5% bone marrow blasts. If studied pretreatment, CR with negativity for a genetic marker by real-time quantitative polymerase chain reaction (RT-qPCR) or similar modality or CR with negativity by multi-color flow cytometry. CR per ELN criteria is defined as neutrophils ≥1.0 × 10^9/L; platelets ≥100 × 10^9/L and <5% bone marrow blasts. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; MRD positive or unknown.
Time Frame: Up to 5 years
Population: Full Analysis Set included participants with AML who received ≥1 dose of magrolimab. As per the pre-specified analysis, this outcome measure was applicable only for the AML cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 87 | 19 | 6 | 1
percentage of participants | 32.2 [22.6 to 43.1] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 97.5]

3. Primary Outcome: CR Rate for Participants With MDS
Description: The CR rate was the percentage of MDS participants who achieved CR per International Working Group (IWG) 2006 criteria. CR per IWG criteria is defined as bone marrow ≤5% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Peripheral blood should have: Hemoglobin (Hgb) ≥11 g/dL, platelets ≥100 × 10^9/L, neutrophils ≥1.0 × 10^9/L and blasts 0%.
Time Frame: Up to 5 years
Population: Full Analysis Set included participants with MDS who received ≥1 dose of magrolimab. As per the pre-specified analysis, this outcome measure was applicable only for the MDS cohorts.
  For the TN MDS Cohort, only participants with higher MDS risk were included for the analyses of this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 17 | 5 | 10 | 9 | 5 | 3
percentage of participants | 37.5 [21.1 to 56.3] | 30.2 [19.2 to 43.0] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8]

4. Primary Outcome: Percentage of Participants With Red Blood Cell (RBC) Transfusion Independence for Participants With Low-Risk MDS
Description: RBC transfusion independence was defined by the lack of RBC transfusions for at least an 8 week consecutive period at any time after starting therapy.
Time Frame: Up to 8 weeks
Population: Full Analysis Set included participants with low-risk MDS who received ≥1 dose of magrolimab. As per the pre-specified analysis, this outcome measure was applicable only for the low risk MDS cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 9 | 5 | 3
percentage of participants | 44.4 [13.7 to 78.8] | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 70.8]

5. Secondary Outcome: Serum Concentration for Magrolimab in TN/U AML and TN MDS Participants
Time Frame: Predose and/or after 1 hour of infusion (duration 3 hours (± 30 minutes) for 1mg/kg; 2 hours for 15 mg/kg, 30 mg/kg and 60 mg/kg) in Cycles (each cycle of 28 days) 1 to 7, 9, 11, 13, 15, on Days 1, 2, 3, 4, 8, 11, 15, 16, 17, 18, 22, EOT, Safety Follow-up
Population: The Pharmacokinetic (PK) Analysis Set included participants in All Enrolled Analysis Set, who took at least 1 dose of magrolimab and had at least 1 detectable postdose magrolimab concentration value reported by the PK laboratory at the given timepoint.
  As per the pre-specified analysis, this outcome measure was applicable only for the TN/U AML and TN MDS cohorts. Data is reported according to the frequency of magrolimab administered: QW, Q2W, QW to Q2W for both TN/U AML and TN MDS cohorts.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- TN/U AML Cohort: Magrolimab + Azacitidine QW: Participants received magrolimab 1 mg/kg on Cycle 1 Days 1 and 4, (C1D1,4) 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15, and 22 and 30 mg/kg QW from Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- TN/U AML Cohort: Magrolimab + Azacitidine Q2W: Participants received magrolimab 1 mg/kg on Cycle 1 Days 1 and 4, (C1D1,4) 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15, and 22 and 30 mg/kg Q2W from Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- TN/U AML Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W; TN MDS Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, 30 mg/kg QW on C2D1, 8, 15 and 22. From Cycle 3 participants received ≥ 1 dose of 30 mg/kg QW and switched to magrolimab 30 mg/kg Q2W.
  Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- TN MDS Cohort: Magrolimab + Azacitidine QW: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15 and 22, and 30 mg/kg QW. From Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- TN MDS Cohort: Magrolimab + Azacitidine Q2W: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15 and 22, and 30mg/kg Q2W from Cycle 3 onwards. Aza was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
Arm/Group | TN/U AML Cohort: Magrolimab + Azacitidine QW | TN/U AML Cohort: Magrolimab + Azacitidine Q2W | TN/U AML Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W | TN MDS Cohort: Magrolimab + Azacitidine QW | TN MDS Cohort: Magrolimab + Azacitidine Q2W | TN MDS Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W
Number analyzed (Participants) | 29 | 42 | 9 | 24 | 56 | 14
ug/mL
  C1D1 Predose: number analyzed (Participants) | 29 | 42 | 9 | 24 | 52 | 13
  C1D1 Predose | 0.18 (0.958) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  C1D1 1 hour: number analyzed (Participants) | 27 | 36 | 6 | 23 | 56 | 12
  C1D1 1 hour | 0.41 (0.830) | 0.29 (0.377) | 0.19 (0.218) | 16.54 (76.838) | 0.40 (0.615) | 0.77 (0.696)
  C1D4 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C1D4 Predose | 0.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C1D4 1 hour: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C1D4 1 hour | 0.32 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C1D8 Predose: number analyzed (Participants) | 27 | 36 | 9 | 23 | 47 | 14
  C1D8 Predose | 0.00 (0.00) | 0.07 (0.398) | 0.00 (0.00) | 17.39 (83.188) | 0.00 (0.00) | 0.00 (0.00)
  C1D8 1 hour: number analyzed (Participants) | 24 | 36 | 7 | 22 | 43 | 13
  C1D8 1 hour | 254.58 (53.242) | 309.17 (103.697) | 258.43 (72.514) | 304.36 (49.765) | 293.09 (75.213) | 262.54 (68.001)
  C1D11 Predose: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 1
  C1D11 Predose | 38.50 (4.384) | 0.00 (0.00) |  | 95.70 (NA) — Standard deviation cannot be calculated for 1 participant. |  | 189.00 (NA) — Standard deviation cannot be calculated for 1 participant.
  C1D11 1 hour: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  C1D11 1 hour | 318.00 (NA) — Standard deviation cannot be calculated for 1 participant. | 338.00 (0.00) |  |  |  |
  C1D15 Predose: number analyzed (Participants) | 24 | 36 | 8 | 18 | 47 | 14
  C1D15 Predose | 320.62 (166.137) | 348.98 (138.719) | 237.01 (109.654) | 360.06 (115.170) | 349.13 (93.294) | 348.64 (142.833)
  C1D15 1 hour: number analyzed (Participants) | 8 | 4 | 1 | 4 | 4 | 1
  C1D15 1 hour | 778.88 (268.194) | 732.50 (335.509) | 578.00 (NA) — Standard deviation cannot be calculated for 1 participant. | 1016.75 (131.801) | 754.00 (207.456) | 887.00 (NA) — Standard deviation cannot be calculated for 1 participant.
  C1D16 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C1D16 Predose | 351.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C1D17 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C1D17 Predose | 278.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C1D18 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C1D18 Predose | 249.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C1D22 Predose: number analyzed (Participants) | 20 | 35 | 8 | 19 | 47 | 14
  C1D22 Predose | 416.80 (131.60) | 374.63 (183.020) | 308.33 (99.219) | 490.05 (151.489) | 437.63 (183.664) | 447.93 (163.772)
  C1D22 1 hour: number analyzed (Participants) | 6 | 4 | 0 | 3 | 3 | 0
  C1D22 1 hour | 873.17 (217.208) | 999.00 (517.850) |  | 1253.33 (123.423) | 790.00 (72.187) |
  C2D1 Predose: number analyzed (Participants) | 20 | 34 | 8 | 20 | 44 | 14
  C2D1 Predose | 398.05 (251.639) | 408.84 (216.656) | 390.50 (104.538) | 480.74 (206.793) | 487.42 (205.862) | 496.57 (179.237)
  C2D1 1 hour: number analyzed (Participants) | 22 | 33 | 8 | 20 | 44 | 11
  C2D1 1 hour | 807.67 (419.553) | 919.33 (313.966) | 948.50 (88.695) | 1009.00 (333.772) | 1078.64 (332.665) | 1064.00 (216.115)
  C2D2 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C2D2 Predose | 0.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C2D3 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C2D3 Predose | 0.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C2D4 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C2D4 Predose | 0.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C2D4 1 hour: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C2D4 1 hour | 1.09 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C2D8 Predose: number analyzed (Participants) | 18 | 35 | 8 | 19 | 39 | 14
  C2D8 Predose | 440.64 (274.761) | 528.31 (244.068) | 458.63 (156.315) | 554.06 (228.605) | 573.62 (213.474) | 491.43 (167.348)
  C2D15 Predose: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0
  C2D15 Predose | 294.00 (213.546) |  |  |  |  |
  C2D22 Predose: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0
  C2D22 Predose | 325.50 (178.898) |  |  |  |  |
  C3D1 Predose: number analyzed (Participants) | 15 | 31 | 8 | 14 | 49 | 13
  C3D1 Predose | 494.00 (222.682) | 549.52 (260.353) | 507.50 (188.883) | 631.87 (216.160) | 597.71 (324.158) | 602.77 (253.499)
  C3D1 1 hour: number analyzed (Participants) | 12 | 27 | 7 | 15 | 40 | 12
  C3D1 1 hour | 971.76 (462.426) | 1245.85 (449.410) | 994.86 (273.703) | 1306.13 (396.321) | 1272.23 (402.487) | 1062.00 (328.337)
  C4D1 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  C4D1 Predose | 336.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |  |  |
  C5D1 Predose: number analyzed (Participants) | 7 | 22 | 8 | 8 | 34 | 11
  C5D1 Predose | 673.29 (183.521) | 301.28 (143.219) | 513.38 (238.555) | 666.38 (317.290) | 246.76 (164.420) | 542.00 (319.484)
  C5D1 1 hour: number analyzed (Participants) | 6 | 21 | 8 | 7 | 33 | 13
  C5D1 1 hour | 1150.50 (342.217) | 1063.43 (445.885) | 1140.78 (343.685) | 1242.99 (691.574) | 917.67 (318.951) | 1104.69 (488.709)
  C6D1 Predose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  C6D1 Predose |  |  |  | 850.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |
  C7D1 Predose: number analyzed (Participants) | 6 | 16 | 9 | 3 | 27 | 10
  C7D1 Predose | 781.83 (256.528) | 274.20 (148.275) | 629.56 (268.028) | 628.00 (504.250) | 281.01 (190.602) | 495.76 (352.143)
  C7D1 1 hour: number analyzed (Participants) | 6 | 14 | 6 | 3 | 25 | 11
  C7D1 1 hour | 1243.17 (344.023) | 932.50 (270.978) | 1297.50 (310.962) | 1325.33 (673.298) | 1007.87 (365.807) | 1039.36 (312.776)
  C9D1 Predose: number analyzed (Participants) | 2 | 7 | 8 | 2 | 19 | 9
  C9D1 Predose | 584.00 (318.198) | 250.71 (122.473) | 522.56 (266.403) | 712.50 (689.429) | 339.06 (170.950) | 401.78 (283.485)
  C9D1 1 hour: number analyzed (Participants) | 2 | 6 | 8 | 2 | 16 | 8
  C9D1 1 hour | 1290.00 (608.112) | 772.50 (296.855) | 1146.88 (304.099) | 1170.50 (635.689) | 1218.19 (245.934) | 1036.63 (313.181)
  C11D1 Predose: number analyzed (Participants) | 0 | 2 | 7 | 0 | 11 | 7
  C11D1 Predose |  | 172.40 (111.157) | 422.29 (315.174) |  | 511.27 (360.621) | 545.81 (332.891)
  C11D1 1 hour: number analyzed (Participants) | 0 | 2 | 8 | 0 | 10 | 6
  C11D1 1 hour |  | 542.50 (365.574) | 988.63 (372.345) |  | 1367.50 (343.182) | 1352.83 (389.004)
  C13D1 Predose: number analyzed (Participants) | 0 | 4 | 5 | 0 | 8 | 6
  C13D1 Predose |  | 349.50 (204.719) | 422.00 (174.360) |  | 370.75 (138.914) | 291.67 (177.293)
  C13D1 1 hour: number analyzed (Participants) | 0 | 4 | 4 | 0 | 8 | 5
  C13D1 1 hour |  | 998.25 (111.870) | 1210.00 (223.756) |  | 1212.88 (531.496) | 968.20 (249.544)
  C15D1 Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  C15D1 Predose |  |  | 443.00 (NA) — Standard deviation cannot be calculated for 1 participant. |  |  |
  End of Treatment (EOT, Up to 4 years): number analyzed (Participants) | 13 | 31 | 5 | 15 | 37 | 8
  End of Treatment (EOT, Up to 4 years) | 298.96 (203.651) | 231.47 (203.912) | 290.82 (138.712) | 611.91 (411.501) | 311.15 (307.602) | 288.39 (184.303)
  Safety Follow-up (FU, Up to 4 years plus 30 days): number analyzed (Participants) | 5 | 14 | 2 | 11 | 21 | 3
  Safety Follow-up (FU, Up to 4 years plus 30 days) | 29.36 (33.138) | 78.26 (90.758) | 152.00 (57.983) | 235.96 (189.895) | 106.45 (198.336) | 32.97 (44.045)

6. Secondary Outcome: Percentage of Participants Who Developed Anti-Magrolimab Antibodies
Description: As per the pre-specified analysis, this outcome measure was analyzed based on different dosing regimens and timepoints when magrolimab was given alone and in combination with the azacitidine. Therefore, the data is reported for magrolimab as monotherapy and magrolimab plus azacitidine. Also, the arms are based on the frequency of magrolimab administered: QW, Q2W, QW to Q2W, Q4W, BIW and BIW to QW as applicable in different cohorts.
Time Frame: Up to 5 years
Population: The Immunogenicity Analysis Set included participants in All Enrolled Analysis Set, who took at least 1 dose of magrolimab and have at least 1 anti-drug antibody (ADA) sample result reported.
Measure: Number; unit: percentage of participants
Groups:
- R/R AML Cohort: Magrolimab + Azacitidine QW: Participants received magrolimab 1 mg/kg on Cycle 1 Days 1 and 4, (C1D1,4) 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15, and 22 and 30 mg/kg QW from Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- R/R AML Cohort: Magrolimab + Azacitidine Q2W: Participants received magrolimab 1 mg/kg on Cycle 1 Days 1 and 4, (C1D1,4) 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15, and 22 and 30 mg/kg Q2W from Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab + Azacitidine QW; TN/U AML Cohort: Magrolimab + Azacitidine QW; TN MDS Cohort: Magrolimab + Azacitidine QW: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15 and 22, and 30 mg/kg QW. From Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab + Azacitidine Q2W: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15 and 22, and 30mg/kg Q2W from Cycle 3 onwards. Azacitidine was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- TN/U AML Cohort: Magrolimab + Azacitidine Q2W; TN MDS Cohort: Magrolimab + Azacitidine Q2W: Participants received magrolimab 1 mg/kg on C1D1, 4, 15 mg/kg on C1D8, 30 mg/kg on C1D11,15 and 22, then 30 mg/kg QW on C2D1, 8, 15 and 22, and 30mg/kg Q2W from Cycle 3 onwards. Aza was given based on approved labeling at standard dose of 75 mg/m^2 on Days 1-7 of each 28-day cycle. Maximum treatment duration was up to 4 years.
- R/R AML Cohort: Magrolimab BIW or BIW to QW: Participants received magrolimab 1 mg/kg on Days 1 and 4, 15 mg/kg on Day 8, and 30 mg/kg on Day 11 and twice weekly (BIW) thereafter for magrolimab monotherapy. From Cycle 3 participants switched from 30 mg/kg BIW to magrolimab 30 mg/kg QW. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab BIW or BIW to QW: Participants received magrolimab 1 mg/kg on Days 1 and 4, 15 mg/kg on Day 8, and 30 mg/kg on Day 11 and twice weekly thereafter for magrolimab monotherapy. From Cycle 3 participants switched from 30 mg/kg BIW to magrolimab 30 mg/kg QW. Maximum treatment duration was up to 4 years.
- R/R MDS Cohort: Magrolimab Q2W: Participants received 1 mg/kg magrolimab on Cycle 1 (Days 1, 4); 15 mg/kg on Cycle 1 Day 8; 30 mg/kg on Cycle 1 Day 11, 15, 22, and then weekly starting Cycle 2 and given as Q2W from Cycle 3 up to end of the study. Maximum treatment duration was up to 4 years.
- Low-Risk MDS Cohort: Magrolimab Q4W: Participants received magrolimab 1 mg/kg on Day 1, 30 mg/kg QW for Cycle 1, followed by 60 mg/kg every 4 weeks (Q4W) from Cycle 2 onward. Maximum treatment duration was up to 4 years.
- Rollover AML Cohort: Magrolimab QW: Dosing schedule may be twice weekly (Day 1, 4, 8, 11, 15, 18, 22, and 25), once weekly (Day 1, 8, 15, 22), or in accordance with a modified recommended Phase 2 dose and schedule determined by the Clinical Trial Steering Committee (CTSC).
  Participants may receive the same dose level and schedule (i.e., twice weekly) of magrolimab monotherapy in each cycle (each cycle was of 28 days) as previously received on the Phase 1 AML study (SCI-CD47-002) or may transition to once-weekly dosing in this study at the discretion of the Investigator in each 28-day cycle and with Sponsor approval. Maximum treatment duration was up to 4 years.
Arm/Group | R/R AML Cohort: Magrolimab + Azacitidine QW | R/R AML Cohort: Magrolimab + Azacitidine Q2W | R/R MDS Cohort: Magrolimab + Azacitidine QW | R/R MDS Cohort: Magrolimab + Azacitidine Q2W | TN/U AML Cohort: Magrolimab + Azacitidine QW | TN/U AML Cohort: Magrolimab + Azacitidine Q2W | TN/U AML Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W | TN MDS Cohort: Magrolimab + Azacitidine QW | TN MDS Cohort: Magrolimab + Azacitidine Q2W | TN MDS Cohort: Magrolimab to Magrolimab + Azacitidine QW to Q2W | R/R AML Cohort: Magrolimab BIW or BIW to QW | R/R MDS Cohort: Magrolimab BIW or BIW to QW | R/R MDS Cohort: Magrolimab Q2W | Low-Risk MDS Cohort: Magrolimab Q4W | Rollover AML Cohort: Magrolimab QW
Number analyzed (Participants) | 9 | 10 | 5 | 12 | 30 | 48 | 9 | 26 | 56 | 14 | 6 | 4 | 11 | 16 | 1
percentage of participants | 0 | 0 | 0 | 0 | 6.7 | 4.7 | 11.1 | 0 | 3.9 | 0 | 16.7 | 0 | 18.2 | 6.7 | 0

7. Secondary Outcome: Duration of Complete Remission (DCR) in Participants With AML and MDS
Description: For AML participants: The DCR was defined as the time measurement criteria were first met for CR (including morphologic CR, CRMRD-, cytogenetic complete remission (cCR), and molecular complete remission (mCR) until the first date that recurrent disease or death with evidence of no disease recurrence was objectively documented. CR and CRMRD- were defined in outcome measure 2. cCR was defined as complete disappearance of chromosomal abnormality without appearance of new ones. mCR was defined as morphological blast of ≤ 5% and recovery of absolute neutrophil count (ANC), platelets, and hemoglobin from complete blood counts as well as peripheral blast.
  For MDS participants: The DCR was defined as the time measurement criteria were first met for CR until the first date that recurrent disease or death with evidence of no disease recurrence is objectively documented.
  Kaplan-Meier (KM) estimates were used in the outcome measure analysis.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set with CR were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included. As per the pre-specified analysis, this outcome measure was applicable only for the all AML and TN MDS cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 12 | 19 | 28 | 0 | 0 | 0
months | 14.4 [3.7 to NA] — Upper limit of confidence interval (CI) was not reached due to insufficient number of events. | 8.5 [7.3 to 12.9] | 9.4 [5.1 to 11.6] |  |  |

8. Secondary Outcome: Percentage of MDS Participants With Objective Response Rate (ORR) as Defined by IWG 2006 MDS Response Criteria
Description: ORR was the percentage of participants who achieved CR, partial remission (PR), marrow CR or hematological improvement (HI) prior to initiation of a new anticancer therapy including SCT per IWG 2006 criteria per investigator's evaluation. CR was defined in outcome measure 2. PR was defined as all CR criteria if abnormal before treatment except the bone marrow blasts decreased by 50% over pretreatment but still > 5% and cellularity and morphology not relevant. Marrow CR is defined as bone marrow ≤5% myeloblasts and decrease by ≥50% over pretreatment, stable disease with any hematological improvement, peripheral blood: if hematological improvement responses, they were noted in addition to marrow CR. Stable Disease: Failure to achieve at least PR, but no evidence of progression for > 8 weeks.
  Percentages were rounded off.
Time Frame: Up to 5 years
Population: Participants with MDS in the Full Analysis Set with data available were analyzed. For the TN MDS Cohort, only participants with higher risk MDS were included. As per the pre-specified analysis, this outcome measure was applicable only the MDS cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 17 | 5 | 10 | 9 | 5 | 3
percentage of participants | 81.3 [63.6 to 92.8] | 69.8 [57.0 to 80.8] | 23.5 [6.8 to 49.9] | 0.0 [0.0 to 52.2] | 10.0 [0.3 to 44.5] | 33.3 [7.5 to 70.1] | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 70.8]

9. Secondary Outcome: Percentage of AML Participants With Objective Response Rate (ORR)
Description: ORR is the percentage of participants who achieve CR, CR with incomplete hematologic (count) recovery (CRi), CR with partial hematologic (count) recovery (CRh), Partial Response (PR), Morphologic Leukemia-Free State (MLFS) prior to initiation of a new anti-cancer therapy including SCT per European Leukemia Net (ELN) AML 2017 recommendations per investigator's evaluation. CR was defined in outcome measure 2. CRi was defined as neutrophils ≥ 1.0 × 10^9/L or platelets ≥ 100 × 10^9/L bone marrow blasts < 5%. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; MRD positive or unknown. CRh was defined in outcome measure 10. PR was defined in outcome measure 8. MLFS was defined as bone marrow blasts < 5%. Absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required; marrow should not merely be "aplastic"; at least 200 cells should be enumerated or cellularity should be at least 10%.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set with AML were analyzed. As per the pre-specified analysis, this outcome measure was applicable only for all AML cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 87 | 19 | 6 | 1
percentage of participants | 47.1 [36.3 to 58.1] | 21.1 [6.1 to 45.6] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 97.5]

10. Secondary Outcome: Percentage of Participants With Complete Remission With Partial Hematologic Recovery (CRh) for AML Participants
Description: CRh was defined as CR with partial platelet and absolute neutrophil count recovery while on study prior to initiation of any new anti-acute myeloid leukemia (AML) therapy or stem cell transplant (SCT).
Time Frame: Up to 5 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 87 | 19 | 6 | 1
percentage of participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Duration of Response (DOR) for Participants With AML
Description: The DOR was defined as time measurement criteria were met for complete remission (CR) (including morphologic CR, CRMRD-, cytogenetic complete remission (cCR), and molecular complete remission (mCR), incomplete blood count recovery (CRi), partial hematologic recovery (CRh), partial remission (PR), marrow CR, or morphologic leukemia-free state (MLFS), whichever was first recorded, until the first date that recurrent or progressive disease, or death with evidence of no disease magrolimab progression is objectively documented. CR and CRMRD- were defined in outcome measure 2. cCR and mCR were defined in outcome measure 7. Marrow CR and PR were defined in outcome measure 8. CRi and MLFS were defined in outcome measure 9. CRh was defined in outcome measure 10.
  KM estimates were used in the outcome measure analysis.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set with AML who achieved ORR were analyzed. As per the pre-specified analysis, this outcome measure was applicable only for the AML cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 41 | 4 | 1 | 1
months | 8.7 [7.4 to 10.4] | 2.7 [0.7 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 2.1 [NA to NA] — Lower and upper limit of CI were not reached due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limit of CI were not reached due to insufficient number of events.

12. Secondary Outcome: Duration of Response for Participants With MDS
Description: The DOR was measured from the time measurement criteria were first met for objective response as assessed by IWG MDS criteria until the first date that recurrent disease or death with evidence of no disease recurrence is objectively documented.
  KM estimates were used in the outcome measure analysis.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set with TN MDS who achieved ORR were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included.
  As per the pre-specified analysis, this outcome measure was applicable for only TN MDS cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg
Number analyzed (Participants) | 26 | 44
months | 12.9 [7.6 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 9.5 [7.9 to 12.9]

13. Secondary Outcome: Overall Survival (OS) for Participants With AML or MDS
Description: The length of overall survival will be measured from the date of study treatment initiation until the date of death from any cause.
  KM estimates were used in the outcome measure analysis.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 87 | 19 | 6 | 1 | 17 | 5 | 10 | 9 | 5 | 3
months | NA [17.7 to NA] — Median and upper limit of CI were not reached due to insufficient number of events. | 19.4 [13.4 to 24.7] | 10.8 [7.2 to 12.8] | 5.2 [1.4 to 9.9] | 8.5 [4.5 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 33.6 [NA to NA] — Lower and upper limit of CI were not reached due to insufficient number of events. | 8.5 [3.7 to 14.7] | 14.1 [7.8 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 4.2 [2.3 to NA] — Upper limit of CI was not reached due to insufficient number of events. | NA [0.6 to NA] — Median and upper limit of CI were not reached due to insufficient number of events. | NA [3.5 to NA] — Median and upper limit of CI were not reached due to insufficient number of events. | 30.6 [30.6 to NA] — Upper limit of CI was not reached due to insufficient number of events.

14. Secondary Outcome: Progression Free Survival (PFS) for Participants With AML or MDS
Description: The length of PFS is defined as the time from the date of study treatment initiation until the date of documented disease progression (PD) or death from any cause, whichever occurs first.
  PD for MDS: <5% blasts: if blasts increase ≥50% to >5%; 5%-10% blasts: if blasts increase ≥50% to >10%; 10%-20% blasts: if blasts increase ≥50% to >20%; 20%-30% blasts: if blasts increase ≥50% to >30%. Participants with at least 50% decrement from maximum remission/response in granulocytes / platelets or reduction in Hgb by ≥ 2 g/dL or transfusion dependence. PD for AML was defined as any evidence for an increase in bone marrow blast percentage and/or increase of absolute blast counts in the blood: > 50% increase in marrow blasts over baseline (a minimum 15% point increase is required in cases with < 30% blasts at baseline; or persistent marrow blast percentage of >70% over at least 3 months; without at least a 100% improvement in absolute neutrophil count.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included.
  As per the pre-specified analysis, this outcome measure was applicable only for all AML and TN MDS cohorts.
  KM estimates were used in the outcome measure analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 87 | 19 | 6 | 1
months | 14.0 [8.6 to 20.4] | 10.7 [7.6 to 11.8] | 7.3 [4.4 to 9.7] | 2.6 [1.0 to 6.0] | 5.2 [0.9 to NA] — Upper limit of CI was not reached due to insufficient number of events. | 1.9 [NA to NA] — Lower and upper limit of CI were not reached due to insufficient number of events.

15. Secondary Outcome: Relapse Free Survival (RFS) for Participants With AML or MDS
Description: The length of RFS is defined from the first date of attaining a CR (including morphologic CR, CRMRD-, cCR, and mCR) until the date of AML relapse or death from any cause, whichever occurs first.
Time Frame: Up to 5 years
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 12 | 19 | 28 | 0 | 0 | 0
months | 14.4 [3.7 to NA] — Upper limit of confidence interval (CI) was not reached due to insufficient number of participants with events. | 8.5 [7.3 to 12.9] | 9.4 [5.1 to 11.6] |  |  |

16. Secondary Outcome: Event Free Survival (EFS) for Participants With AML or MDS
Description: For AML, EFS was defined as the time from the date of study treatment initiation until the date of documented disease progression, death from any cause, or treatment failure (defined as failure to achieve CR/CRi/CRh by Cycle 5 Day 1), whichever occurred first. CR/CRi/CRh were defined in outcome measures 2, 9 and 10 respectively.
  For MDS, EFS was defined as the time from the date of study treatment initiation to transformation to AML or death from any cause, whichever occurred first. Participants who were not observed to have one of these events during the study were censored at their last response assessment date with evidence of no transformation to AML.
  KM estimates were used in the outcome measure analysis.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included.
  As per the pre-specified analysis, this outcome measure was applicable only for all AML and TN MDS cohorts.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 87 | 19 | 6 | 1
months | 18.2 [12.9 to NA] — Upper limit of CI were not reached due to insufficient number of events. | 23.1 [11.8 to NA] — Upper limit of CI were not reached due to insufficient number of events. | 3.7 [2.1 to 7.3] | 1.7 [0.8 to 3.5] | 1.4 [0.0 to NA] — Upper limit of CI were not reached due to insufficient number of events. | 1.9 [NA to NA] — Lower and upper limit of CI were not reached due to insufficient number of events.

17. Secondary Outcome: Change From Baseline in Hemoglobin on Therapy
Time Frame: Baseline and Day 1
Population: Participants in the Safety Analysis Set were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included. As per the pre-specified analysis, this outcome measure was applicable only for the R/R AML and TN MDS cohorts.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN MDS Cohort Low Risk QW 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 1 | 87 | 19 | 6 | 1
g/dL
  Baseline | 8.5 (1.56) | 9.0 (1.50) | 10.1 (NA) — Standard deviation cannot be calculated for 1 participant. | 8.8 (1.27) | 9.1 (1.39) | 10.3 (1.74) | 8.9 (NA) — Standard deviation cannot be calculated for 1 participant.
  Change at Day 1: number analyzed (Participants) | 31 | 61 | 1 | 84 | 19 | 6 | 1
  Change at Day 1 | -0.1 (1.23) | -0.7 (1.10) | -0.7 (NA) — Standard deviation cannot be calculated for 1 participant. | -0.8 (1.08) | -0.9 (0.92) | -1.3 (1.32) | 0.1 (NA) — Standard deviation cannot be calculated for 1 participant.

18. Secondary Outcome: 12-week RBC Transfusion Independence Rates
Time Frame: Up to 12 Weeks
Population: Data was not collected for this outcome measure.
Arm/Group | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Minimal Residual Disease (MRD) Negative Response Rate
Description: The MRD-negative response rate was defined as the percentage of participants who reach MRD-negative disease status prior to initiation of other new anti-cancer therapy including SCT and achieve a morphologic CR or marrow CR for MDS participants and achieve CR/CRi/CRh/MLFS for AML participants. MRD-negative disease status will be assessed using a multiparameter flow cytometry-based assay performed by a central laboratory. CR/CRi/MLFS/CRh were defined in outcome measures 2, 9, 10 respectively. Marrow CR was defined in outcome measure 8.
Time Frame: Up to 5 years
Population: Participants in the Full Analysis Set with MDS were analyzed. For the TN MDS Cohort, only participants with higher MDS risk were included.
  As per the pre-specified analysis, this outcome measure was applicable only for all AML and TN MDS cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab
Number analyzed (Participants) | 32 | 63 | 87 | 19 | 6 | 1
percentage of participants | 28.1 [13.7 to 46.7] | 20.6 [11.5 to 32.7] | 21.8 [13.7 to 32.0] | 5.3 [0.1 to 26.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 97.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 5 years; Adverse events: Up to 4 years
Description: All-cause mortality: All Enrolled Analysis Set included all participants who were enrolled into the study.
  Adverse events: Safety Analysis Set included all participants who received ≥ 1 dose of magrolimab.
Arm/Group | TN MDS Cohort Higher Risk QW 30 mg/kg | TN MDS Cohort Higher Risk Q2W 30 mg/kg | TN MDS Cohort Low Risk QW 30 mg/kg | TN/U AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab + Azacitidine | R/R AML Cohort: Magrolimab | Rollover AML Cohort: Magrolimab | R/R MDS Cohort: Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine | R/R MDS Cohort: Magrolimab | Low Risk MDS Cohort: Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine | Low Risk MDS Cohort: Magrolimab
All-Cause Mortality (participants affected / at risk) | 12/32 | 44/63 | 1/1 | 72/87 | 18/19 | 6/6 | 1/1 | 15/17 | 3/5 | 7/10 | 3/9 | 1/5 | 1/3
Serious Adverse Events (participants affected / at risk) | 20/32 | 40/63 | 0/1 | 64/87 | 17/19 | 4/6 | 1/1 | 12/17 | 2/5 | 7/10 | 8/9 | 3/5 | 1/3
Other Adverse Events (participants affected / at risk) | 32/32 | 60/63 | 1/1 | 84/87 | 19/19 | 6/6 | 1/1 | 17/17 | 5/5 | 10/10 | 9/9 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TN MDS Cohort Higher Risk QW 30 mg/kg (N=32) | TN MDS Cohort Higher Risk Q2W 30 mg/kg (N=63) | TN MDS Cohort Low Risk QW 30 mg/kg (N=1) | TN/U AML Cohort: Magrolimab + Azacitidine (N=87) | R/R AML Cohort: Magrolimab + Azacitidine (N=19) | R/R AML Cohort: Magrolimab (N=6) | Rollover AML Cohort: Magrolimab (N=1) | R/R MDS Cohort: Magrolimab + Azacitidine (N=17) | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine (N=5) | R/R MDS Cohort: Magrolimab (N=10) | Low Risk MDS Cohort: Magrolimab + Azacitidine (N=9) | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine (N=5) | Low Risk MDS Cohort: Magrolimab (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 16 | 0 | 21 | 6 | 2 | 1 | 4 | 1 | 2 | 1 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell agglutination (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 6 | 0 | 4 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 6 | 0 | 11 | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 2 | 1 | 0 | 1 | 5 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 6 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sars-cov-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal amyloidosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TN MDS Cohort Higher Risk QW 30 mg/kg (N=32) | TN MDS Cohort Higher Risk Q2W 30 mg/kg (N=63) | TN MDS Cohort Low Risk QW 30 mg/kg (N=1) | TN/U AML Cohort: Magrolimab + Azacitidine (N=87) | R/R AML Cohort: Magrolimab + Azacitidine (N=19) | R/R AML Cohort: Magrolimab (N=6) | Rollover AML Cohort: Magrolimab (N=1) | R/R MDS Cohort: Magrolimab + Azacitidine (N=17) | R/R MDS Cohort: Magrolimab to Magrolimab + Azacitidine (N=5) | R/R MDS Cohort: Magrolimab (N=10) | Low Risk MDS Cohort: Magrolimab + Azacitidine (N=9) | Low Risk MDS Cohort: Magrolimab to Magrolimab + Azacitidine (N=5) | Low Risk MDS Cohort: Magrolimab (N=3)
Anaemia (Blood and lymphatic system disorders) | 15 | 31 | 0 | 30 | 1 | 2 | 1 | 8 | 3 | 4 | 4 | 4 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 0 | 23 | 8 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 9 | 1 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Red blood cell agglutination (Blood and lymphatic system disorders) | 3 | 2 | 1 | 6 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 9 | 0 | 14 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 2 | 0 | 8 | 3 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 4 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 14 | 0 | 20 | 4 | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 26 | 40 | 1 | 43 | 9 | 2 | 0 | 9 | 2 | 2 | 4 | 4 | 1
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 27 | 0 | 42 | 9 | 1 | 0 | 6 | 2 | 2 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 0 | 7 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 0 | 11 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 0 | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 5 | 0 | 7 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 33 | 1 | 42 | 7 | 1 | 0 | 9 | 2 | 2 | 5 | 0 | 1
Oral blood blister (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 5 | 0 | 5 | 4 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 17 | 1 | 21 | 4 | 1 | 0 | 6 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 8 | 0 | 8 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Catheter site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 3 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 6 | 14 | 0 | 19 | 3 | 0 | 0 | 6 | 3 | 0 | 1 | 0 | 1
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 15 | 20 | 0 | 34 | 4 | 1 | 0 | 6 | 2 | 3 | 4 | 1 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 3 | 4 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 3 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 6 | 15 | 0 | 26 | 5 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 3 | 0 | 4 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 11 | 11 | 0 | 26 | 3 | 0 | 0 | 5 | 1 | 2 | 1 | 1 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0 | 7 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Device related bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 3 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 0 | 7 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 5 | 0 | 7 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Vaginal cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 9 | 0 | 9 | 2 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 12 | 0 | 22 | 5 | 2 | 0 | 5 | 0 | 1 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 15 | 0 | 15 | 3 | 0 | 0 | 8 | 1 | 3 | 4 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 5 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 8 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 6 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 12 | 0 | 17 | 4 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 12 | 0 | 13 | 5 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 0 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 11 | 23 | 1 | 20 | 4 | 1 | 0 | 4 | 0 | 2 | 3 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 6 | 6 | 0 | 3 | 3 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haptoglobin decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 3 | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Klebsiella test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 17 | 19 | 0 | 15 | 3 | 0 | 0 | 3 | 1 | 1 | 3 | 2 | 0
Platelet count decreased (Investigations) | 14 | 27 | 0 | 24 | 2 | 1 | 0 | 6 | 2 | 1 | 4 | 3 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 5 | 9 | 0 | 13 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 15 | 15 | 0 | 14 | 3 | 0 | 0 | 3 | 1 | 1 | 2 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 22 | 0 | 29 | 4 | 0 | 0 | 3 | 0 | 2 | 3 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 6 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 8 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 9 | 4 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 4 | 6 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 15 | 1 | 23 | 9 | 1 | 0 | 6 | 0 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 7 | 0 | 9 | 4 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 8 | 1 | 15 | 5 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 11 | 1 | 22 | 8 | 0 | 0 | 7 | 1 | 0 | 0 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 0 | 14 | 5 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 0 | 11 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Deep tissue injury (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 11 | 2 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 5 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 4 | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 10 | 0 | 13 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 16 | 0 | 24 | 4 | 2 | 0 | 3 | 0 | 1 | 4 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 7 | 0 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 22 | 1 | 21 | 6 | 1 | 0 | 4 | 0 | 1 | 2 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vith nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 0 | 10 | 4 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 4 | 1 | 0 | 11 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 9 | 0 | 14 | 4 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 0 | 10 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 3 | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 3 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 16 | 0 | 28 | 7 | 3 | 0 | 7 | 1 | 2 | 3 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 22 | 1 | 21 | 6 | 1 | 0 | 7 | 1 | 3 | 3 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 17 | 6 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 11 | 4 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 9 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oropharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 9 | 4 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 10 | 2 | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 5 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 13 | 0 | 10 | 5 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 7 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 9 | 0 | 10 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 6 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 8 | 5 | 1 | 6 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 7 | 8 | 0 | 17 | 7 | 1 | 0 | 4 | 1 | 3 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03248479/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT03248479/SAP_001.pdf